CLINICAL TRIAL: NCT00488813
Title: Association of Antibiotic Utilization Measures and Control of Extended-spectrum β-lactamases (ESBLs) in MICU1 and MICU2 at Buddhist Tzu Chi General Hospital.
Brief Title: Study of Antibiotic Utilization Measures and Control of ESBLs in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101441
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: ICU Patient
Keywords: Tzh-Chi ESBL study
MeSH Terms: interventions — Third Generation Cephalosporins

INTERVENTIONS:
Drug: Third generation cephalosporins

SUMMARY:
A single-center, prospective, comparative, antibiotic intervention study for patients admitted to MICU1 and MICU2

DETAILED DESCRIPTION:
1. To determine the value of using β-lactamases inhibitors in reducing the cases of ESBL producing E. coli or K. pneumoniae colonization and infection after 12 months.
2. To compare the acquisition rates of ESBL producing E. coli or K. pneumoniae at MICU1 and MICU2 after 12 months

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted or transferred to the ICU/burn units.
* Patients of either sex, 18 years of age or older.

Exclusion Criteria:

* Patient with hypersensitivity to penicillins, cephalosporins, and beta-lactamase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
For both MICU1 and MICU2 (acquisition), all culture results will be collected and recorded, then analyzed to determine the ESBL acquisition rate and bacterial isolates (E. coli or K. pneumoniae).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com